CLINICAL TRIAL: NCT04270071
Title: Efficacy and Safety of Yangxin Shengmai Granules for the Treatment of Stable Angina Pectoris: Randomised, Double Blind, Placebo Controlled Trial
Brief Title: Efficacy and Safety of Yangxin Shengmai Granules for the Treatment of Stable Angina Pectoris
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Jun Li, Chief physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YXSM_2019001
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Coronary Heart Disease; Stable Angina
Keywords: Yangxinshengmai granules; Stable angina pectoris; Coronary heart disease; Randomized controlled trial
MeSH Terms: conditions — Coronary Disease; Angina, Stable | interventions — Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yangxin Shengmai Granules (Experimental): Patients were given Yangxin Shengmai granules orally 14g (1 bag) each time, 3 times daily for 4 weeks. And nitroglycerin tablets are used when angina attack.
  For patients who have used drugs such as aspirin, angiotensin-converting enzyme inhibitor, lipid-lowering drugs to treat coronary heart disease before inclusion, they can continue to use the original varieties and doses, without dose adjustment.
  Interventions: Drug: Yangxin Shengmai; Drug: nitroglycerin tablets
- Placebo (Placebo Comparator): Patients were given Yangxin Shengmai granules simulation orally 14g (1 bag) each time, 3 times daily for 4 weeks. And nitroglycerin tablets are used when angina attack.
  For patients who have used drugs such as aspirin, angiotensin-converting enzyme inhibitor, lipid-lowering drugs to treat coronary heart disease before inclusion, they can continue to use the original varieties and doses, without dose adjustment.
  Interventions: Drug: Yangxin Shengmai placebo; Drug: nitroglycerin tablets

INTERVENTIONS:
Drug: Yangxin Shengmai — Yangxin Shengmai Granules
  Other Names: YXSM
  Arms: Yangxin Shengmai Granules
Drug: Yangxin Shengmai placebo — Yangxin Shengmai placebo have an identical appearance and scent as the active treatment granules.
  Other Names: YXSM placebo
  Arms: Placebo
Drug: nitroglycerin tablets — Be used when angina attack

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, parallel clinical trial in Chinese population with stable angina pectoris. The purpose is to determine the efficacy and safety of Yangxin Shengmai Granules in the treatment of stable angina pectoris.

DETAILED DESCRIPTION:
Yangxin Shengmai granules is a Chinese patent medicine composed of ginseng, Ophiopogon japonicus, Salvia miltiorrhiza, Schisandra chinensis, etc. It is used for the treatment of chest pain caused by Qi-yin deficiency and blood stasis in traditional Chinese medicine. The symptoms include chest tightness, chest pain, palpitation, shortness of breath, fatigue, dry mouth and dry throat. Clinical applications suggested that Yangxin Shengmai granules were safe and effective in the treatment of coronary heart disease. However, high-quality clinical trials are still needed to further confirm, so as to provide theoretical basis for the treatment of stable angina pectoris with traditional Chinese medicine.

The study is designed to determine the efficacy and safety of Yangxin Shengmai Granules in the treatment of stable angina pectoris.

ELIGIBILITY:
Inclusion Criteria:

* Participants are aged between 40 and 75 years.
* Meet the diagnostic criteria of stable angina pectoris.
* Meet Chinese medicine syndrome differentiation of Qi-yin deficiency and blood stasis syndrome.
* Voluntarily participate and sign informed consent.

Exclusion Criteria:

* Patients were diagnosed as acute myocardial infarction, unstable angina, stable exertion angina and other heart diseases.
* Patients with poor control of hypertension and diabetes, severe cardiopulmonary insufficiency, severe arrhythmia (rapid atrial fibrillation, atrial flutter, paroxysmal ventricular tachycardia, etc.), with a history of heart pacemaker or cerebrovascular disease within one year.
* Any of the following disease history or evidence was found in the screening period: severe cardiovascular or cerebrovascular diseases; active, recurrent peptic ulcer or other bleeding risk diseases; other serious diseases of digestive system; combined with malignant tumor, blood system disease, serious or progressive diseases of the other system; combined with mental diseases.
* Before screening, any laboratory inspection index meets the following standards: The results showed that Glutamic aspartate transaminase (AST) or alanine aminotransferase (ALT) were more than 1.5 times of the upper limit of normal value and serum creatinine (Cr) was more than 1.2 times of the upper limit of normal value.
* With a history of alcohol and drug abuse.
* Pregnant or lactating women.
* Patients who have participated in clinical trials of other drugs within 3 months before enrollment.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Stopping or reducing rate of the nitroglycerin tablets | Four weeks after treatment
  Number of nitroglycerin tablets used before medication - number of nitroglycerin tablets used after medication) / number of nitroglycerin tablets used before medication × 100%

SECONDARY OUTCOMES:
Changes of angina symptom score | Two and four weeks after treatment
  The angina symptom score regroups three items: degree of the frequency, duration and severity of angina attacks. The score of each item is 0,2,4,6. And higher scores mean a worse outcome.
Patient-reported outcomes in coronary heart disease | Two and four weeks after treatment
  Through clinical outcome evaluation scale for patients with coronary heart disease with angina pectoris

CONTACTS AND LOCATIONS:
Overall Officials: Jun Li, MD, Study Director — Guang'anmen Hospital of China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu S, Tian G, Chen J, Zhang X, Wu A, Li M, Sun Y, Liu B, Xing Y, Shang H. Traditional Chinese Medicine for Bradyarrhythmia: Evidence and Potential Mechanisms. Front Pharmacol. 2018 Apr 9;9:324. doi: 10.3389/fphar.2018.00324. eCollection 2018. PMID 29686614
- [Result] Walters MA. Management of Chronic Stable Angina. Crit Care Nurs Clin North Am. 2017 Dec;29(4):487-493. doi: 10.1016/j.cnc.2017.08.008. Epub 2017 Sep 29. PMID 29107310
- [Result] Kallistratos MS, Poulimenos LE, Manolis AJ. Beta blockers, calcium channel blockers, and long-acting nitrates for patients with stable angina and low blood pressure levels: should this recommendation be reconsidered? Eur Heart J. 2020 Jan 14;41(3):479. doi: 10.1093/eurheartj/ehz900. No abstract available. PMID 31883335
- [Result] Chen M, Men L, Wu H, Zhong G, Ou L, Li T, Guo Y, Lin H, Zhang J, Wang D, Zhang Z. A systematic review of the effectiveness and safety of Chinese herbal medicine formula Gualou Xiebai Banxia (GLXBBX) decoction for the treatment of stable angina pectoris. Medicine (Baltimore). 2019 Dec;98(51):e18375. doi: 10.1097/MD.0000000000018375. PMID 31860998
- [Result] Li Y, Zhang L, Lv S, Wang X, Zhang J, Tian X, Zhang Y, Chen B, Liu D, Yang J, Dong P, Xu Y, Song Y, Shi J, Li L, Wang X, Han Y. Efficacy and safety of oral Guanxinshutong capsules in patients with stable angina pectoris in China: a prospective, multicenter, double-blind, placebo-controlled, randomized clinical trial. BMC Complement Altern Med. 2019 Dec 11;19(1):363. doi: 10.1186/s12906-019-2778-z. PMID 31829173
- [Result] Surveillance report 2016 - Stable angina: management (2011) NICE guideline CG126 [Internet]. London: National Institute for Health and Care Excellence (NICE); 2016 Apr 3. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK551066/ PMID 31855330
- [Result] Yang X, He T, Han S, Zhang X, Sun Y, Xing Y, Shang H. The Role of Traditional Chinese Medicine in the Regulation of Oxidative Stress in Treating Coronary Heart Disease. Oxid Med Cell Longev. 2019 Feb 24;2019:3231424. doi: 10.1155/2019/3231424. eCollection 2019. PMID 30918578
- [Result] Gong P, Li Y, Yao C, Guo H, Hwang H, Liu X, Xu Y, Wang X. Traditional Chinese Medicine on the Treatment of Coronary Heart Disease in Recent 20 Years. J Altern Complement Med. 2017 Sep;23(9):659-666. doi: 10.1089/acm.2016.0420. Epub 2017 May 12. PMID 28497986
- [Result] Li GH, Jiang HY, Xie YM, Jiang JJ, Yang W, Zhao W, Zhuang Y, Wang YY. [Analysis of traditional Chinese medicine syndrome, traditional Chinese medicine and western medicine in 84 697 patients with coronary heart disease based on big data]. Zhongguo Zhong Yao Za Zhi. 2014 Sep;39(18):3462-8. Chinese. PMID 25532378